CLINICAL TRIAL: NCT01364064
Title: Conventional Adjuvant Temozolomide With Dose Intensive Temozolomide in Patients With Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Collaborators: Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAC#2081-018
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2013-09

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional adjuvant Temozolomide (Active Comparator): TMZ d 1-5 of 28-d cycle 6 cycles
  Interventions: Drug: TMZ
- Dose intensive Temozolomide (Experimental): TMZ d 1-21 of 28-d cycle 6 cycles
  Interventions: Drug: TMZ

INTERVENTIONS:
Drug: TMZ — Comparing conventional adjuvant Temozolomide with dose intensive Temozolomide

SUMMARY:
This is a Phase III Trial Comparing Conventional Adjuvant Temozolomide with Dose Intensive Temozolomide in Patients with Newly Diagnosed Glioblastoma.

DETAILED DESCRIPTION:
Primary objective is to determine if dose-intensifying (increasing the "dose-density") the adjuvant temozolomide component of the chemoradiation treatment enhances treatment efficacy as measured by overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Karnofsky performance status of ≥ 60. 2. Age ≥ 18 years. 4. CBC/differential obtained within 14 days prior to study registration, with adequate bone marrow function as defined below:

* Absolute neutrophil count (ANC) ≥ 1500 cells/mm3.
* Platelets ≥ 100,000 cells/mm3.
* Hemoglobin ≥ 10 g/dl. (Note: The use of transfusion or other intervention to achieve Hgb ≥ 10 g/dl is acceptable.)
* Adequate renal function, as defined below:
* BUN ≤ 25 mg/dl within 14 days prior to study registration
* Creatinine ≤ 1.7 mg/dl within 14 days prior to study registration 4. Adequate hepatic function, as defined below:
* Bilirubin ≤ 2.0 mg/dl within 14 days prior to study registration
* ALT ≤ 3 x normal range within 14 days prior to study registration
* AST ≤ 3 x normal range within 14 days prior to study registration 5. Patients must sign a study-specific informed consent prior to study registration.

If the patient's mental status precludes his/her giving informed consent, written informed consent may be given by the responsible family member.

6. For females of child-bearing potential, negative serum pregnancy test within 72 hours prior to starting temozolomide.

7. Women of childbearing potential and male participants must practice adequate contraception.

Exclusion Criteria:

1. Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for ≥ 3 years. (For example, carcinoma in situ of the breast, oral cavity, and cervix are all permissible).
2. Recurrent or multifocal malignant gliomas
3. Metastases detected below the tentorium or beyond the cranial vault.
4. Prior chemotherapy or radiosensitizers for cancers of the head and neck region; note that prior chemotherapy for a different cancer is allowable. Prior use of Gliadel wafers or any other intratumoral or intracavitary treatment are not permitted.
5. Prior radiotherapy to the head or neck (except for T1 glottic cancer), resulting in overlap of radiation fields.
6. Severe, active co-morbidity, defined as follows:

   * Unstable angina and/or congestive heart failure requiring hospitalization
   * Transmural myocardial infarction within the last 6 months
   * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
   * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
   * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol.
   * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
   * Major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy.
   * Active connective tissue disorders, such as lupus or scleroderma, that in the opinion of the treating physician may put the patient at high risk for radiation toxicity.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1153 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
safety and efficacy | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Naseer Al-Rajhi, Principal Investigator — KFSH & RC